CLINICAL TRIAL: NCT07373821
Title: Influence of Supine Positioning on the Outcomes After Descemet Membrane Endothelial Keratoplasty (DMEK)
Acronym: SUPINE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Maximilian Friedrich, Principal Investigator, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-400/2025
Record Dates: First submitted 2025-10-02; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Fuchs Endothelial Corneal Dystrophy; Descemet Membrane Endothelial Keratoplasty (DMEK)
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 day supine positioning (Experimental)
  Interventions: Procedure: Duration of Supine Positioning
- 5 day supine positioning (Active Comparator)
  Interventions: Procedure: Duration of Supine Positioning

INTERVENTIONS:
Procedure: Duration of Supine Positioning — 1 day supine positioning vs 5 days supine positioning

SUMMARY:
The goal of this clinical trial is to learn if a longer period of lying on the back after corneal transplant surgery (Descemet Membrane Endothelial Keratoplasty, DMEK) helps the transplant stick better in the eye. It will also learn about side effects, such as back pain.

The main questions it aims to answer are:

* Does lying on the back for 5 days reduce the size of transplant detachment compared to lying on the back for only 1 day?
* Do participants who lie on their back longer need fewer additional procedures (rebubbling)?
* What symptoms or problems do participants experience with short vs. long back positioning?

Researchers will compare two groups:

* 1 day of back positioning
* 5 days of back positioning

Participants will:

* Be randomly assigned to one of the two positioning groups
* Wear a movement sensor that records head position
* Have their eyes checked regularly with vision tests and imaging (AS-OCT)
* Answer questions about their vision and comfort
* Keep a diary of any positioning-related complaints, such as back pain

ELIGIBILITY:
Inclusion Criteria:

Fuchs Endothelial Corneal Dystrophy Bullous Keratopathy

Exclusion Criteria:

Comorbidities preventing supine positioning

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Area of Graft Detachment in mm² | First two postoperative weeks
  The area of graft detachment will be measured in mm² using anterior segment optical coherence tomography and a custom-built segmentation tool

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, University Hospital Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No